CLINICAL TRIAL: NCT04445935
Title: Anticoagulation in Patients Suffering From COVID-19 Disease-The Anti-Co Trial
Brief Title: Anticoagulation in Patients Suffering From COVID-19 Disease The ANTI-CO Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Marcus Daniel Lance, Professor Dr. Marcus Lance, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MRC-05-082
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Anticoagulation in COVID-19 ARDS
Keywords: COVID-19; ARDS; Anticoagulation
MeSH Terms: conditions — COVID-19 | interventions — bivalirudin

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will be blinded to the above mentioned group. The PI is not involved in active treatment. Patients are sedated and ventilated when treatment starts and finally the outcome assessors will not be knowing the patients treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment (Active Comparator): In this arm the patients will be treated according to our standard anticoagulation protocol.
  The patients will not be treated with Bivalirudin (the investigational drug).
  Interventions: Drug: Standard treatment
- Bivalirudin arm (Experimental): The patients will be anticoagulated according to the institutional HIT-protocol which uses Bivalirudin as anticoagulant.
  Interventions: Drug: Bivalirudin Injection

INTERVENTIONS:
Drug: Bivalirudin Injection — The patients will receive iv Bivalirudin according to the institutional HIT protocol.
  Other Names: anticoagulation
  Arms: Bivalirudin arm
Drug: Standard treatment — This group will receive standard anticoagulation with LMWH/UFH
  Arms: Standard treatment

SUMMARY:
Patients with COVID-19 associated ARDS and mechanical ventilation have a high mortality. Part of the disease is an activation of the coagulation system which seems to contribute to clotformation in the pulmonary bloodstream. Recently we implemented an algorithm applying higher doses of heparins (LMWH). However, this approach could not inhibit clotformation enough. Bivalirudin could prevent clotformation better and support dissolving existing clots.

Therefore, we want to compare 50 patients with the standard treatment with 50 patients under bivalirudin treatment which we normally apply in patients with a HIT-syndrome.

Our primary outcome measure is oxygenation reflected as P/F ratio.

DETAILED DESCRIPTION:
The pandemic of COVID-19, a newly upcoming viral disease caused by SARS-CoV-2, puts the whole worlds health system under pressure.

Patients suffering from this disease mainly develop respiratory symptoms, which can lead to severe acute respiratory distress syndrome (ARDS) necessitating ICU admission in 10-20% of the cases admitted to hospital. In addition to these symptoms, patients show lymphopenia, cardiac symptoms and altered coagulation profiles. Although those patients are treated in the ICU the mortality there is more than 20% due to multiorgan failure.

One of the recent insights in this disease is its effect on the coagulation system. Meanwhile we know that the coagulation system gets activated. Furthermore, it seems that clot formation takes place in the pulmonary micro-vasculature which could contribute to the widely observed gas-exchange impairment. Therefore, many centers apply empiric anticoagulation for their COVID-patients. At the moment, we at HMC, also apply an empirical anticoagulation protocol as our standard approach. However, this is a symptomatic treatment without good proof.

Bivalirudin is a well-known agent which is used in HMC for cases in which anticoagulation is needed, but a contraindication for heparin exists (i.e. HIT syndrome). This drug has an interesting pharmacologic profile. It acts independent of antithrombin (AT), the physiological compound which enhances heparin effects under normal circumstances. This lack of dependence on AT, makes Bivalirudin an attractive choice in light of the contradictory reports on the levels of AT during COVID infection. If AT levels are decreased during the infection, heparin (as well as LMWH) cannot work efficiently, which would render our treatment less effective. Luckily, bivalirudin acts without the support of AT, so we could bypass this problem. In addition, bivalirudin has some fibrinolytic activities. It inhibits clot-bound thrombin which as a result destabilizes the clot rendering it more susceptible to thrombolysis. This property partially supports the dissolving of clots and could support re-opening the pulmonary microcirculation.

Objectives:

To prove the positive effect of anticoagulation with bivalirudin intravenously on gas-exchange in patients with COVID-19 and respiratory failure on invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years of age)
* Positive COVID-test
* Under mechanical ventilation
* D-Dimers>1.2 mg/L

Exclusion Criteria:

* Pregnancy
* Allergy to the drug (bivalirudin)
* Inherited coagulation abnormalities
* No informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-28 (Estimated); Primary Completion 2020-09-28 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
P/F ratio | three days of intervention
  the P/F ratio is a surrogate parameter for oxygenation in ARDS.

SECONDARY OUTCOMES:
Kidney function | three days of intervention
  The kidney function frequently is deteriorated in COVID-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lance, MD, PhD, Principal Investigator — HMC
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
this will depend on IRB advice

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Kharma N, Roehrig S, Shible AA, Elshafei MS, Osman D, Elsaid IM, Mustafa SF, Aldabi A, Smain OAM, Lance MD. Anticoagulation in critically ill patients on mechanical ventilation suffering from COVID-19 disease, The ANTI-CO trial: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Sep 7;21(1):769. doi: 10.1186/s13063-020-04689-1. PMID 32895056